CLINICAL TRIAL: NCT05295160
Title: Fasting-Associated Immune-metabolic Remission of Diabetes Type 2
Brief Title: Fasting-Associated Immune-metabolic Remission of Diabetes
Acronym: FAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Senior Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAIR-EFSD
Record Dates: First submitted 2020-09-25; First posted 2022-03-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: type 2 diabetes mellitus in obese; insulin secretion; innate immunity; monocyte programming; remission of type 2 diabetes; weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Obese people with type 2 diabetes with a duration of less then 4 years will be compared with people with type 2 diabetes for more than 8 years regarding their capability to achieve remission of type 2 diabetes in response to a weight loss of 15kg achived using very low calorie intake
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- type 2 diabetes - less than 4 years duration (Other): Patients with a duration of less than 4 years since diagnosis of type 2 diabetes, BMI > 28 kg/m², non-insulin treated who agree to loose 15 kg body weight by eating a very low calorie formula diet of 800 kcal/day for men and 600 kcal/day for women. The duration of the diet is until the weight loss is achieved.
  Interventions: Behavioral: weight loss by very low energy diet intake which may differ in protein or carbohydrate content
- type 2 diabetes - more than 8 years (Other): Patients with a duration of more than 8 years since diagnosis of type 2 diabetes, BMI > 28 kg/m², non-insulin treated who agree to loose 15 kg body weight by eating a very low calorie formula diet of 800 kcal/day for men and 600 kcal/day for women. The duration of the diet is until the weight loss is achieved.
  Interventions: Behavioral: weight loss by very low energy diet intake which may differ in protein or carbohydrate content

INTERVENTIONS:
Behavioral: weight loss by very low energy diet intake which may differ in protein or carbohydrate content — The anthropometric, endocrine and metabolic status is tested before, after 7 days and after 15 kg weight loss

SUMMARY:
People with a body mass index above 28 kg/m² and an onset of type 2 diabetes within the last 4 years had a remission (HbA1c <6.5% without medication) of diabetes in over 80% upon weight loss of 15 kg. Longer duration of diabetes reduced the chance of remission. The investigators will test whether there is a difference in remission upon weight loss of 15 kg using formula low calorie diets between subjects with a diabetes duration of <4 years vs. >8 years and oral treatment as primary end points. The immune metabolic programming of circulating monocytes will be investigated in detail regarding trained innate immunity and the endocrine responses will be determined using meal challenge tests.

DETAILED DESCRIPTION:
A remission of type 2 diabetes can be achieved in over 80% of people with a diagnosis within the last 4 years and overweight or obesity by weight loss of 15 kg. The mechanisms involve an improvement of insulin sensitivity and thereby insulin requirements and a regain of the function of insulin secreting beta cells. Longer duration of type 2 diabetes appears to impair the capacity of beta cell to regenerate. At present it is not possibe to predict success of the weight loss at an early time point. The investigators therefore aim to identify early markers of responders. It is unclear how the weight loss induces the remission in responders. Immune cells are known to contribute to insulin resistance by regulating adipose tissue function and hepatic and skeletal muscle metabolism by releasing cytokines. The inborn immune system is known to adapt to external stimuli by the process of trained immunity and is thought to contribute to insulin resistance and the dysfunction of beta-cells. The investigation will analyze the programming state of innate immune cells in detail in the course of diabetes remission. In addition, islet hormone responses to challenge tests will be performed to assess their function in detail.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed less than 4 or over 8 years, before study,
* BMI > 28 kg/m²,
* willingness to follow weight loss diet,

Exclusion Criteria:

* consuming disease,
* intolerance for very low calorie formula diet,
* known severe hepatic disease or liver cirrhosis,
* type 1 diabetes,
* severe disease of kidney or heart,
* advanced diabetic retinopathy,
* intake of glucocorticoids,
* drug or alcohol abuse,
* weight loss of >5 kg in the last 3 month,
* eating disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Concentration of fasting blood glucose < 126 mg/deciliter | 3 month
  Remission of type 2 diabetes defined by a concentration of a fasting blood glucose < 126 mg/deciliter without diabetes medication

SECONDARY OUTCOMES:
Immune-metabolic profile and programing of innate immunity | before, after 7 days and after 3 month
  Changes of cluster of differentiation 4/cluster of differentiation antigen 45 circulating immune cells in percent of CD4+ cells measured by flow cytometry in blood.
  Concentrations of TNFalpha in pg/ml, changes of Momocyte Chemoattractant Protein-1 in pg/ml.
Composition of the microbiome | before, after 7 days and after 3 month
  Percent changes in firmicutes in stool,

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, MD, Study Director — Universitätsmedizin Berlin CBF
Locations (1):
- Charité Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Steven S, Hollingsworth KG, Al-Mrabeh A, Avery L, Aribisala B, Caslake M, Taylor R. Very Low-Calorie Diet and 6 Months of Weight Stability in Type 2 Diabetes: Pathophysiological Changes in Responders and Nonresponders. Diabetes Care. 2016 May;39(5):808-15. doi: 10.2337/dc15-1942. Epub 2016 Mar 21. PMID 27002059